CLINICAL TRIAL: NCT03660956
Title: Comparative Effects of Exercise and Back Counselling on Improving Low Back Pain for Nurses
Brief Title: Effects of Exercise and Back Counselling for Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CMUH107-REC2-120
Record Dates: First submitted 2018-08-30; First posted 2018-09-07 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A Quasi-Experimental design is used in this study. Participants are randomly assigned to exercise and back counselling group or back counselling only group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise and back counselling group (Experimental)
  Interventions: Behavioral: Exercise; Behavioral: Back counselling
- Back counselling group (Active Comparator)
  Interventions: Behavioral: Back counselling

INTERVENTIONS:
Behavioral: Exercise — Twelves-week exercise training sessions include a variety of strength, flexibility, and coordination exercises. Each exercise session lasts for one hour. Participants are expected to attend exercise session once a week and are encouraged to continue exercising at home.
  Arms: Exercise and back counselling group
Behavioral: Back counselling — Procedure of back counselling includes one session back counselling, lasting one hour. The topics of back counselling session are as follows: (1) Anatomy of lumbar; (2) Factors causing low back pain; (3) Problems of physical inactivity for the lumbar; (4) Risk of poor postures for developing persistent/chronic low back pain; (5) Maintaining right posture of the lumbar; (6) Avoiding harmful loading of the back during work and leisure time.

SUMMARY:
Low back pain (LBP) is most common occupational health problem among nurses. Therefore, how to prevent and reduce low back pain have been the important issue for nurses. A Quasi-Experimental design is used in this study to compare the effectiveness of 12-week exercise and counselling program to reduce low back pain in nursing personnel compared with counselling alone.

DETAILED DESCRIPTION:
A Quasi-Experimental design is used in this study. Purposive sampling is used to recruit participants from medical center in Central Taiwan. Participants will be randomly assigned to two groups: (1) exercise and back counselling, and (2) back counselling only. The results of this study will provide a guideline for nurses to prevent and to improve low back pain.

ELIGIBILITY:
Inclusion Criteria:

1. Has worked at current job for at least 12 months;
2. Intensity of low back pain on Visual Analogue Scale (scale 0-10) at least two during the past 3 months.

Exclusion Criteria:

1. Serious former back injury (fracture, surgery, disc protrusion);
2. Pregnant;
3. Other serious disease or symptoms that limit participation exercise defined by a physician.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Pain on Visual Analogue Scale (VAS) at week 6, week 12, month 3, and month 6 | Baseline, week 6, week 12, month 3, month 6.
  Visual Analogue Scale (VAS) is used in this study to assess the intensity of low back pain with numeric rating scale 0-100 mm during the past month.

SECONDARY OUTCOMES:
Change from Baseline Musculoskeletal Symptoms in the Low Back Area at week 6, week 12, month 3 and month 6 | Baseline, week 6, week 12, month 3, month 6.
  Version of the low back questionnaire in Nordic Musculoskeletal Questionnaire (NMQ) is used in this study to assess the musculoskeletal symptoms in the low back area.
Change from Baseline Functional Status at week 6, week 12, month 3 and month 6 | Baseline, week 6, week 12, month 3, month 6
  Chinese version of Oswestry Disability Index (ODI) is used in this study to assess the baseline functional status and its change over time for patients with back pain

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Hsin Shih, PhD, Principal Investigator — China Medical University, China
Locations (1):
- China Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No